CLINICAL TRIAL: NCT04017598
Title: Is Iron Supplementation Harmful in Populations Where Iron Deficiency is Not the Cause of Anemia? A 12 Week Randomized Controlled Trial in Cambodia
Brief Title: Potential Harms of Untargeted Iron Supplementation in Cambodia Where Iron Deficiency is Not the Cause of Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Helen Keller International (Other); NCHADS - Ministry of Health of Cambodia (Other); BC Children's Hospital Research Institute (Other); The National Institute of Public Health Laboratory, Phnom Penh (Unknown)
Responsible Party: Principal Investigator, Crystal Karakochuk, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H18-02610
Record Dates: First submitted 2019-07-04; First posted 2019-07-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Anemia, Iron Deficiency; Anemia; Intestinal Inflammation; Inflammation; Intestine; Complaints
Keywords: anemia; gut inflammation; iron deficiency; iron; iron supplementation
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Inflammation; Iron Deficiencies | interventions — ferrous sulfate; Iron-Dextran Complex; ferrous bisglycinate; iron(III) N,N'-bis((5-bromo-2-hydroxyphenyl)glycinate); Salts

STUDY DESIGN:
Intervention Model Description: 12-week double-blind, three-arm, placebo-controlled randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The manufacturers of the tablets (Dr. Simon Wood, Natural Factors) will be responsible for allocation concealment of the three tablet formulations at time of packaging. All tablets will be non-distinguishable in size, colour, and packaging. Trial investigators, research staff, and participants will all be blinded to the assigned interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ferrous Sulfate (Active Comparator): Iron will be given orally in the form of tablets. A supplement of 60 mg will be taken daily for 12 weeks. World Health Organization standard dose and commonly used form of iron.
  Interventions: Dietary Supplement: Ferrous sulfate
- Ferrous Bisglycinate (Experimental): Iron will be given orally in the form of tablets. A supplement of 18 mg will be taken daily for 12 weeks. Ferrous bisglycinate has a bioavailability 2-4x greater than ferrous sulfate.
  Interventions: Dietary Supplement: Ferrous Bisglycinate
- Placebo (Placebo Comparator): Placebo will be given orally in the form of tablets as a control made of microcrystalline cellulose.
  Interventions: Dietary Supplement: Placebo of microcrystalline cellulose

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — 60 mg elemental iron as ferrous sulfate
  Other Names: iron sulfate; ferrous sulphate; iron sulphate; Iron(II) sulfate
  Arms: Ferrous Sulfate
Dietary Supplement: Ferrous Bisglycinate — 18 mg elemental iron as ferrous bisglycinate
  Other Names: iron amino acid chelate; Iron glycinate; Bisglycine iron(II) salt; Iron(II) bisglycinate; Ferrous Bis-glycinate
  Arms: Ferrous Bisglycinate
Dietary Supplement: Placebo of microcrystalline cellulose — placebo
  Other Names: Control
  Arms: Placebo

SUMMARY:
In 2016, the World Health Organization (WHO) set a global policy recommending daily oral iron supplementation (60 mg iron) for 12 weeks for all women living in countries where anemia prevalence is >40%, such as in Cambodia. However, recent studies have shown the prevalence of iron deficiency to be low in Cambodian women and that supplementation would likely only benefit ~10% of women.

Iron supplementation may be harmful in women with genetic blood disorders (e.g. thalassemia), which are common in Cambodia, as these individuals are already at an increased risk of iron overload. The risks are made greater by the fact that iron absorption from most common form of supplementation, ferrous sulfate, is low. Typically less than 20% is absorbed in the gut; the remaining 80% passes unabsorbed into the colon where it can increase the risk of pathogen growth and gut inflammation. Alternatively, ferrous bisglycinate is a newer supplemental form of iron. This amino acid chelate has 2-4x higher bioavailability than ferrous sulfate and is associated with fewer GI side-effects.

In view of WHO policy and risks of supplementation, there is a need to determine the potential for harm, and if novel forms of iron supplements are safer.

DETAILED DESCRIPTION:
The World Health Organization (WHO) set a Global Nutrition Target to reduce anemia in women of reproductive age by 50% by 2025. In 2016, the WHO implemented a global policy recommending oral iron supplementation (60 mg daily for 12 weeks) for all women where anemia prevalence is more than 40%, such as in Cambodia.

However, recent studies have shown the prevalence of iron deficiency to be low in Cambodian women. If iron deficiency is not the cause of anemia, then iron supplementation will not be effective at treating it. Further, iron supplementation may be harmful in some individuals, especially those with anemia caused by genetic blood disorders (which are common in Cambodia), as these individuals are already at an increased risk of iron overload. The risks are made greater by the fact that the type of iron that is commonly used in supplements (ferrous sulfate) is poorly absorbed. Typically, less than 20% is absorbed in the gut; the remaining 80% is unabsorbed in the colon where it can increase the risk of pathogen growth and gut inflammation.

To investigate the safety of untargeted iron supplementation, we will undertake a new study in Cambodia, where we will evaluate a newer type of iron supplement that may be absorbed better, and thus, safer than the conventional type. We will recruit non-pregnant women (18-45 years) and ask them to take one of the two forms of iron (ferrous sulfate or ferrous bisglycinate) or a placebo for 12 weeks (in line with the WHO global policy). We will measure hemoglobin and ferritin levels, which are markers of anemia and iron status, and markers of gut inflammation and gut pathogen abundance, before and after the intervention. This study will contribute to the evidence for safe and effective iron supplementation for women worldwide.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy
* consent to participate in the study and provide blood, flocked rectal swab and stool samples
* expected to reside in the study location for the study period.

Exclusion Criteria:

* any known illness or disease
* pregnant
* taking antibiotics, non-steroidal anti-inflammatory drugs, dietary supplements, or vitamin and mineral supplements in the previous 12 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 480 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Serum Ferritin | 12 weeks
  Serum ferritin concentration (µg/l) at 12 weeks
Fecal calprotectin | 12 weeks
  Fecal calprotectin concentration (mg/kg stool) at 12 weeks as a measure of gut inflammation.

SECONDARY OUTCOMES:
Gut pathogen abundance | 12 weeks
  Real-time PCR nucleic acid amplification assay with an enteric bacterial panel.
Gut parasite abundance | 12 weeks
  Real-time PCR nucleic acid amplification assay with an enteric parasite panel.
DNA damage | 12 weeks
  DNA damage will be assessed by measuring DNA single-strand breaks, indicated by olive tail movement with use of alkali single-cell gel electrophoresis (Comet assay).
Alpha-1 acid glycoprotein (AGP, g/l) | 12 weeks
C-reactive protein (CRP, mg/l) | 12 weeks
Hemoglobin (g/L) | 12 weeks
Folate (ng/ml) | 12 weeks
Vitamin B12 (pmol/l) | 12 weeks

OTHER OUTCOMES:
Reported side effects | Continuous over 12 weeks
  (e.g., gastrointestinal pain) as a quality of life measure.
Genetic hemoglobinopathies | Baseline
  Genotyping to detect the presence of the most common hemoglobinopathies
Gut Pathogen abundance | 12 weeks
  Whole metagenome shotgun 16S ribosomal RNA sequencing will be conducted on fecal samples, in order to validate the method against the established BD MAX panel in a subset of 150 women from our trial (50 from each study arm).

CONTACTS AND LOCATIONS:
Locations (1):
- Prey Kuy, Srayov and Tboung Krapeu Health Centres, Kampong Thom, Cambodia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Cirigliano E, Saint A, Pei LX, Wong CW, Wang S, Fischer JA, Kroeun H, Karakochuk CD. Iron Supplementation with Ferrous Sulfate or Ferrous Bisglycinate for 12 Weeks Does Not Influence Group B Streptococcus Colonization in Cambodian Women: A Secondary Analysis of a Randomized Controlled Trial. J Nutr. 2025 Dec;155(12):4264-4270. doi: 10.1016/j.tjnut.2025.10.014. Epub 2025 Oct 11. PMID 41082982
- [Derived] Fischer JAJ, Pei LX, Elango R, Hou K, Goldfarb DM, Karakochuk CD. Is a Lower Dose of More Bioavailable Iron (18-mg Ferrous Bisglycinate) Noninferior to 60-mg Ferrous Sulfate in Increasing Ferritin Concentrations While Reducing Gut Inflammation and Enteropathogen Detection in Cambodian Women? A Randomized Controlled Noninferiority Trial. J Nutr. 2023 Aug;153(8):2453-2462. doi: 10.1016/j.tjnut.2023.05.029. Epub 2023 Jun 2. PMID 37271416
- [Derived] Finlayson-Trick E, Nearing J, Fischer JA, Ma Y, Wang S, Krouen H, Goldfarb DM, Karakochuk CD. The Effect of Oral Iron Supplementation on Gut Microbial Composition: a Secondary Analysis of a Double-Blind, Randomized Controlled Trial among Cambodian Women of Reproductive Age. Microbiol Spectr. 2023 Jun 15;11(3):e0527322. doi: 10.1128/spectrum.05273-22. Epub 2023 May 18. PMID 37199608
- [Derived] Fischer JA, Pei LX, Goldfarb DM, Albert A, Elango R, Kroeun H, Karakochuk CD. Is untargeted iron supplementation harmful when iron deficiency is not the major cause of anaemia? Study protocol for a double-blind, randomised controlled trial among non-pregnant Cambodian women. BMJ Open. 2020 Aug 16;10(8):e037232. doi: 10.1136/bmjopen-2020-037232. PMID 32801202